CLINICAL TRIAL: NCT00270153
Title: The Use of ACE Inhibitors in the Early Renal Post-transplant Period
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-12-311
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Renal Transplant
Keywords: renal transplant, ACE inhibitor
MeSH Terms: interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- enalapril (Placebo Comparator)
  Interventions: Drug: enalapril
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: enalapril — 5mg enalapril daily for 6 months
  Arms: enalapril
Drug: Placebo — 5mg enalapril-matching placebo daily for 6 months
  Arms: Placebo

SUMMARY:
Chronic allograft nephropathy (CAN) is the leading cause of longterm renal transplant loss. Angiotensin-II may play a role in the development and progression of CAN. Angiotensin converting enzyme inhibitors (ACEI) comprise a drug class that inhibit the effects of angiotensin-II. However these drugs have been reported to cause elevated potassium and creatinine levels in some renal transplant patients. Yet, there are now several retrospective reports of long term benefits of improved renal function and graft survival in renal transplant recipients. There have been no reports of prospective randomized controlled trials of ACEI in renal transplant patients in the early post transplant period.

The purpose of the present study is to assess the safety of enalapril, a drug in the ACEI class, when started 1-3 month post transplant. This is a double-blinded, randomized control trial of enalapril vs. placebo in new renal transplant patients with serum creatinine values no higher than 2.5mg/dl and normal serum potassium levels. The study drug will be administered for 6 months. Patients will be monitored in the renal transplant clinic every 1-4 weeks according to routine protocol. Clinical end-points will be occurence of potassium >5.9mEQ/L or sustained increase in serum creatinine >30% from baseline.

DETAILED DESCRIPTION:
All new renal transplant recipients with functioning allografts and serum creatinine less than 2.6 mg/dl within the first 3 month post transplant would be eligible for this study of the safety of enalapril 5 mg vs placebo. Patients with serum potassium persistently over 5.5 mEQ/L would be excluded. This is a double-blinded randomized control study. End-points of the study are a persistent rise in serum creatinine of >30% from baseline not otherwise explained by clinical evaluation, and persistent serum potassium >5.9mEQ/L. Study duration is 6 month. At the end of the study patients will be continued on ACEI if clinically stable

ELIGIBILITY:
Inclusion Criteria:

* New adult renal transplant recipients with good renal function defined as serum creatinine less than 2.6 mg/dl,
* Normal serum potassium levels,
* No contraindication to ACE inhibitor use

Exclusion Criteria:

* Renal transplant patients with persistent serum creatinine levels over 2.5 mg/dl
* Hyperkalemia with serum potassium levels over 5.5 mEQ/dl
* History of allergic reaction to ACE inhibitors or angiotensin receptor blockers
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in serum creatinine levels assessed at 6 months | Baseline and 6 months
  Creatinine is a waste product that comes from the normal wear and tear on muscles of the body. It is excreted through the kidneys. High serum creatinine levels in the blood indicate that the kidneys aren't functioning properly. Increase in serum creatinine of 30% would be a safety concern and requires clinical management.
Changes in potassium levels assessed at 6 months | Baseline and 6 months
  Potassium is a chemical that is critical to the function of nerve and muscle cells, including those in your heart. Potassium levels must be kept within a very narrow concentration range. High Potassium levels are a sign of worsening kidney function. An occurence of serum potassium greater than 5.9 mEq/L is a safety concern and requires clinical management.
Decrease in estimated glomerular filtration rate (eGFR) assessed at 6 months | Baseline and 6 months.
  eGFR is a number based on your blood test for creatinine, a waste product in your blood.It tells how well your kidneys are working. A normal eGFR is 60 or more. A 25 percent decrease in eGFR indicates that the kidneys may not be working well. This is a safety concern and requires clinical management.

SECONDARY OUTCOMES:
Cough due to drug intolerance assessed at 6 months | Baseline and 6 months
  Cough experienced because of inability to tolerate the adverse effects of the medication
abdominal pain due to drug intolerance assessed at 6 months | Baseline and 6 months
  Abdominal pain experienced because of inability to tolerate the adverse effects of the medication
Erythrocytosis assessed at 6 months | Baseline and 6 months
  Erythrocytosis is a condition in which your body makes too many red blood cells (RBCs). Too many red blood cells can make your blood thicker than normal and lead to blood clots and other complications.
Leukopenia assessed at 6 months | Baseline and 6 months
  Leukopenia is a decrease in the number of white blood cells found in the blood, which places individuals at increased risk of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Coco, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471